CLINICAL TRIAL: NCT00978471
Title: Efficacy and Tolerance Adjuvant High-Dose Thiotepa With Peripheral Stem Cell Rescue Associated With Conventional Chemotherapy in Children and Adults With Relapsed Osteosarcoma
Brief Title: Adjuvant High-Dose Thiotepa and Stem Cell Rescue Associated With Conventional Chemotherapy in Relapsed Osteosarcoma
Acronym: OSII-TTP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSII-TTP; 2009-009899-12 (EudraCT Number)
Record Dates: First submitted 2009-09-16; First posted 2009-09-17 (Estimated); Last update posted 2019-05-17 (Actual); Status verified 2018-08

CONDITIONS: Osteosarcoma
Keywords: Conventional chemotherapy; cytapheresis; Peripheral stem cell autograft; Surgical resection; Thiotepa
MeSH Terms: conditions — Osteosarcoma | interventions — Thiotepa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- experimental arm thiotepa (Experimental): 4 courses of conventional chemotherapy followed by high-dose Thiotepa with peripheral stem cell rescue. Surgical resection of all tumor masses will be performed as soon as possible.
  Interventions: Drug: Thiotepa
- Reference arm (Other): 4 courses of conventional chemotherapy. Surgical resection of all tumor masses will be performed as soon as possible.
  Interventions: Drug: Thiotepa

INTERVENTIONS:
Drug: Thiotepa — Thiotepa 8-12mg/m²/day/injection Total dose for one cure:15-50mg.
  Other Names: N N'N'triethylenethiophosphosphoramide; Tepadina

SUMMARY:
Approximately 150 new cases of osteosarcoma are reported each year in France, of which 15 to 20% are metastatic.

Further to the initial standard care, about 45% of the patients relapse within a median duration of 20 months.

Result of the OS94 study results and of the investigation performed within the CRLCC, indicate that 25 to 30 patients (children and adults) experience an osteosarcoma relapse each year in FRANCE.

According to several studies, the 5-year overall survival rate of patients in first relapse is 23-28%,with a median post relapse survival of 10 to 17 months. Multiple relapse cases are also reported in the COSS study, with a median time to second relapse of 0.8 year.

At present, there is no reference treatment for the standard care of osteosarcoma relapse in FRANCE.

Thiotepa is known for its antitumor effect in numerous malignant tumors. In 2007, a study from our institution reported that about 35% of all osteosarcoma relapses are treated with a high-dose thiotepa while the efficacy and tolerance of this therapeutic strategy have never been assessed.

These results highlight the need to the evaluate the efficacy and tolerance of this high-dose of thiotepa within a clinical trial and its inclusion in the standard care of the osteosarcoma at relapse.

DETAILED DESCRIPTION:
Despite the absence of tumor registry, approximately 150 new cases of osteosarcoma are reported each year in France (100 cases per year in children and 50 cases in adults), of which 15 to 20% are metastatic. The standardized impact rate in the world population is estimated at 3 per million inhabitants per year.

Further to the initial standard care, about 45% of the patients relapse within a median interval of 20 months (range 3 months - 10 years).

Results of the OS94 study and of the investigation performed within the CRLCC indicate that 25 to 30 patients (children and adults) experience an osteosarcoma relapse each year in FRANCE.

Results of the five major published series indicate that the 5-year overall survival rate of patients in first relapse is between 23 and 28%, with a median post-relapse survival of 10 to 17 months. Multiple relapse cases are also reported in the COSS study, with a median time to second relapse of 0.8 year.

At present, there is no reference treatment for the standard care of osteosarcoma relapse in FRANCE.

Some recommendations have been given in the OS94 protocol, but they are generally not followed or they are implemented in a heterogeneous manner.

Thiotepa (N N' N'' triethylenethiophosphoramide), an alkylating agent of the chemical family of ethylene-imines, is known for its antitumor effect in a number of malignant tumors.

Its efficacy in osteosarcoma has been reported in the literature. A retrospective study of the SFCE (French Society for Childhood Cancer, results not yet published) in 45 patients presenting with refractory osteosarcoma or relapse has shown a radiological reaction rate of 30%.

Moreover, a preliminary investigation performed by the CLB in 2007 within the framework of the SFCE study explored all relapse cases diagnosed between the beginning of 2004 and the end of 2006. Results showed that about 35% of the patients with osteosarcoma relapses are treated with high-dose thiotepa while the efficacy and tolerance of this therapeutic strategy have never been assessed.

Altogether, these results led the SFCE osteosarcoma group to propose the evaluation of the efficacy and tolerance of this high-dose thiotepa chemotherapy within a clinical trial and to include the drug in the standard care of osteosarcoma in relapse.

ELIGIBILITY:
Inclusion Criteria:

* Age > 1 year and < 50 years
* First osteosarcoma relapse, either local or metastatic, or second relapse after exclusive surgery NB: Whenever possible, only patients with histological evidence of relapse will be included.
* Indication for chemotherapy confirmed by a multidisciplinary committee.
* Surgical resection of all tumor sites must be possible, either as first-line therapy or after chemotherapy.
* Lansky score ≥ 60%, or ECOG Performance Status ≤ 2
* ≥ 21-day interval after first-line chemotherapy
* Blood tests, renal and liver functions within the normal range for age with, in particular, 7 days prior to study entry, blood or serum values as follows:
* blood: neutrophil count > 1 G/L; platelets >100 G/L
* renal: serum creatinine ≤ 1.5 x ULN depending on age; patients with serum creatinine values > 1.5 x ULN are eligible if creatinine clearance is > 70 mL/min/1.73 m²
* liver: total bilirubin < 2 x ULN; ASAT and ALAT ≤ 5 x ULN
* cardiac: isotopic or echographic Left Ventricular Ejection Fraction > 50 %.
* Signed written informed consent; for children, signed consent from the patient (depending on age) and from the parents or legal representative is mandatory
* Documented negative serum βHCG for female patients of childbearing age
* Affiliation with health insurance.

Exclusion Criteria:

* Patients with multiple relapses for whom surgical resection seems impossible, even after chemotherapy.
* Patients already treated with high-dose chemotherapy regimens
* Patients with a contra-indication to the treatment proposed
* Patients not eligible for leukapheresis
* Two-year follow-up impossible due to social, family, geographic or psychological reasons
* Patient included in another protocol of clinical research
* Pregnant or lactating women.

Ages: 1 Year to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2009-07; Primary Completion 2018-10-29 (Actual); Study Completion 2018-10-29 (Actual)

PRIMARY OUTCOMES:
Estimate the overall survival rate | 24 months

SECONDARY OUTCOMES:
Estimate overall survival after relapse diagnosis | 24 months
Estimate the survival free progression after randomization | 24 months
Evaluate the tolerance profile of experimental treatment (hematologic toxicity) | every 3 weeks
Estimate the rate of tumor response to treatment as assessed by conventional CT-scan | at inclusion, day 14-day 21 after the 2nd chemotherapy cycle, before randomization, day 14-day 21 after the 4th chemotherapy cycle, after thiotepa cure and 8 weeks after the end of treatment
Estimate histological response to treatment on surgical tumor samples | If surgery is applicable, a few weeks after thiotepa cure (12 to 17 weeks after inclusion)
Study of biological and genomic properties and analysis of angiogenic markers correlated with relapse (optional) | At inclusion,at surgery , and at the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Perrine MAREC-BÉRARD, Dr, Principal Investigator — Institut d'Hématologie et d'Oncologie Pédiatrique (IHOP) - CLB
Locations (23):
- France (23):
  - CHU Besançon- Hôpital Jean Minjoz, Besançon
  - Chu - Hopital Des Enfants Bordeaux, Bordeaux
  - CHU Dijon Le Bocage, Hôpital d'Enfants, Dijon
  - Chu Grenoble, Grenoble
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard - Institut d'Hémato-Oncologie Pediatrique, Lyon
  - Institut Paoli Calmettes, Marseille
  - Hôpital des Enfants de la Timone, Marseille
  - Chu Nantes - Hopital Meres Et Enfants, Nantes
  - Centre Antoine Lacassagne, Nice
  - CHU Nice, Hôpital L'Archet 2, Nice
  - Institut Curie, Paris
  - Hopital D'Enfants Armand Trousseau, Paris
  - CHU Poitiers, site de la Milétrie, Poitiers
  - CHU RENNES - Hôpital Sud, Rennes
  - Chu La Reunion, Saint-Denis
  - Institut de Cancérologie de l'Ouest - René Gauducheau, Saint-Herblain
  - CHU de SAINT-ETIENNE, Hôpital Nord, Saint-Priest-en-Jarez
  - Institut Lucien Neurwith, Saint-Priest-en-Jarez
  - Hopital de Hautepierre, Strasbourg
  - Chu Toulouse - Hopital D'Enfants, Toulouse
  - Chu Nancy - Hopital D'Enfants, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Background] Desandes E, Lacour B, Sommelet D, Buemi A, Danzon A, Delafosse P, Grosclaude P, Mace-Lesech J, Raverdy-Bourdon N, Tretarre B, Velten M, Brugieres L. Cancer incidence among adolescents in France. Pediatr Blood Cancer. 2004 Dec;43(7):742-8. doi: 10.1002/pbc.20106. PMID 15390305
- [Background] Widhe B, Widhe T. Initial symptoms and clinical features in osteosarcoma and Ewing sarcoma. J Bone Joint Surg Am. 2000 May;82(5):667-74. doi: 10.2106/00004623-200005000-00007. PMID 10819277
- [Background] Jaffe N, Paed D, Farber S, Traggis D, Geiser C, Kim BS, Das L, Frauenberger G, Djerassi I, Cassady JR. Favorable response of metastatic osteogenic sarcoma to pulse high-dose methotrexate with citrovorum rescue and radiation therapy. Cancer. 1973 Jun;31(6):1367-73. doi: 10.1002/1097-0142(197306)31:63.0.co;2-6. No abstract available. PMID 4541163
- [Background] Gasparini M, Rouesse J, van Oosterom A, Wagener T, Somers R, Russel JA, Voute PA, Bramwell V, Thomas D, Sylvester R, et al. Phase II study of cisplatin in advanced osteogenic sarcoma. European Organization for Research on Treatment of Cancer Soft Tissue and Bone Sarcoma Group. Cancer Treat Rep. 1985 Feb;69(2):211-3. PMID 3855699
- [Background] Marti C, Kroner T, Remagen W, Berchtold W, Cserhati M, Varini M. High-dose ifosfamide in advanced osteosarcoma. Cancer Treat Rep. 1985 Jan;69(1):115-7. PMID 3855382
- [Background] Cores EP, Holland JF, Wang JJ, Sinks LF. Doxorubicin in disseminated osteosarcoma. JAMA. 1972 Sep 4;221(10):1132-8. doi: 10.1001/jama.221.10.1132. No abstract available. PMID 4512088
- [Background] Rosen G, Caparros B, Huvos AG, Kosloff C, Nirenberg A, Cacavio A, Marcove RC, Lane JM, Mehta B, Urban C. Preoperative chemotherapy for osteogenic sarcoma: selection of postoperative adjuvant chemotherapy based on the response of the primary tumor to preoperative chemotherapy. Cancer. 1982 Mar 15;49(6):1221-30. doi: 10.1002/1097-0142(19820315)49:63.0.co;2-e. PMID 6174200
- [Background] Bielack SS, Kempf-Bielack B, Delling G, Exner GU, Flege S, Helmke K, Kotz R, Salzer-Kuntschik M, Werner M, Winkelmann W, Zoubek A, Jurgens H, Winkler K. Prognostic factors in high-grade osteosarcoma of the extremities or trunk: an analysis of 1,702 patients treated on neoadjuvant cooperative osteosarcoma study group protocols. J Clin Oncol. 2002 Feb 1;20(3):776-90. doi: 10.1200/JCO.2002.20.3.776. PMID 11821461
- [Background] Souhami RL, Craft AW, Van der Eijken JW, Nooij M, Spooner D, Bramwell VH, Wierzbicki R, Malcolm AJ, Kirkpatrick A, Uscinska BM, Van Glabbeke M, Machin D. Randomised trial of two regimens of chemotherapy in operable osteosarcoma: a study of the European Osteosarcoma Intergroup. Lancet. 1997 Sep 27;350(9082):911-7. doi: 10.1016/S0140-6736(97)02307-6. PMID 9314869
- [Background] Claude L, Rousmans S, Carrie C, Breteau N, Dijoud F, Gentet JC, Giammarile F, Jouve JL, Kind M, Marec-Berard P, Mascard E, Bataillard A, Philip T; Institut National du Cancer; Fedeation nationale des centres de lutte contre le cancer (FNCLCC); Standards, Options et Recommendations; Ligue nationale contre le cancer; SFCE; Fedeation hospitaliere de France; FNCHRU; Fedeation francaise de cancerologie. [Standards and Options for the use of radiation therapy in the management of patients with osteosarcoma. Update 2004]. Bull Cancer. 2005 Oct;92(10):891-906. French. PMID 16266873
- [Background] Franzius C, Schuck A, Bielack SS. High-dose samarium-153 ethylene diamine tetramethylene phosphonate: low toxicity of skeletal irradiation in patients with osteosarcoma and bone metastases. J Clin Oncol. 2002 Apr 1;20(7):1953-4. doi: 10.1200/JCO.2002.20.7.1953. No abstract available. PMID 11919261
- [Background] Harris MB, Gieser P, Goorin AM, Ayala A, Shochat SJ, Ferguson WS, Holbrook T, Link MP. Treatment of metastatic osteosarcoma at diagnosis: a Pediatric Oncology Group Study. J Clin Oncol. 1998 Nov;16(11):3641-8. doi: 10.1200/JCO.1998.16.11.3641. PMID 9817286
- [Background] Mialou V, Philip T, Kalifa C, Perol D, Gentet JC, Marec-Berard P, Pacquement H, Chastagner P, Defaschelles AS, Hartmann O. Metastatic osteosarcoma at diagnosis: prognostic factors and long-term outcome--the French pediatric experience. Cancer. 2005 Sep 1;104(5):1100-9. doi: 10.1002/cncr.21263. PMID 16015627
- [Background] Crompton BD, Goldsby RE, Weinberg VK, Feren R, O'Donnell RJ, Ablin AR. Survival after recurrence of osteosarcoma: a 20-year experience at a single institution. Pediatr Blood Cancer. 2006 Sep;47(3):255-9. doi: 10.1002/pbc.20580. PMID 16123980
- [Background] Ferrari S, Briccoli A, Mercuri M, Bertoni F, Cesari M, Longhi A, Bacci G. Late relapse in osteosarcoma. J Pediatr Hematol Oncol. 2006 Jul;28(7):418-22. doi: 10.1097/01.mph.0000212944.82361.1d. PMID 16825986
- [Background] Shi XB, Chen AM, Cai XH, Guo FJ, Liao GN, Ma D. Establishment and characterization of cell sublines with high and low metastatic potential derived from human osteosarcoma. Chin Med J (Engl). 2005 Apr 20;118(8):687-90. No abstract available. PMID 15899125
- [Background] Bacci G, Briccoli A, Longhi A, Ferrari S, Mercuri M, Faggioli F, Versari M, Picci P. Treatment and outcome of recurrent osteosarcoma: experience at Rizzoli in 235 patients initially treated with neoadjuvant chemotherapy. Acta Oncol. 2005;44(7):748-55. doi: 10.1080/02841860500327503. PMID 16227167
- [Background] Ferrari S, Briccoli A, Mercuri M, Bertoni F, Picci P, Tienghi A, Del Prever AB, Fagioli F, Comandone A, Bacci G. Postrelapse survival in osteosarcoma of the extremities: prognostic factors for long-term survival. J Clin Oncol. 2003 Feb 15;21(4):710-5. doi: 10.1200/JCO.2003.03.141. PMID 12586810
- [Background] Huth JF, Eilber FR. Patterns of recurrence after resection of osteosarcoma of the extremity. Strategies for treatment of metastases. Arch Surg. 1989 Jan;124(1):122-6. doi: 10.1001/archsurg.1989.01410010132026. PMID 2910240
- [Background] Kempf-Bielack B, Bielack SS, Jurgens H, Branscheid D, Berdel WE, Exner GU, Gobel U, Helmke K, Jundt G, Kabisch H, Kevric M, Klingebiel T, Kotz R, Maas R, Schwarz R, Semik M, Treuner J, Zoubek A, Winkler K. Osteosarcoma relapse after combined modality therapy: an analysis of unselected patients in the Cooperative Osteosarcoma Study Group (COSS). J Clin Oncol. 2005 Jan 20;23(3):559-68. doi: 10.1200/JCO.2005.04.063. PMID 15659502
- [Background] Saeter G, Hoie J, Stenwig AE, Johansson AK, Hannisdal E, Solheim OP. Systemic relapse of patients with osteogenic sarcoma. Prognostic factors for long term survival. Cancer. 1995 Mar 1;75(5):1084-93. doi: 10.1002/1097-0142(19950301)75:53.0.co;2-f. PMID 7850705
- [Background] Tabone MD, Kalifa C, Rodary C, Raquin M, Valteau-Couanet D, Lemerle J. Osteosarcoma recurrences in pediatric patients previously treated with intensive chemotherapy. J Clin Oncol. 1994 Dec;12(12):2614-20. doi: 10.1200/JCO.1994.12.12.2614. PMID 7989936
- [Background] Jeffree GM, Price CH, Sissons HA. The metastatic patterns of osteosarcoma. Br J Cancer. 1975 Jul;32(1):87-107. doi: 10.1038/bjc.1975.136. PMID 1058038
- [Background] Weeden S, Grimer RJ, Cannon SR, Taminiau AH, Uscinska BM; European Osteosarcoma Intergroup. The effect of local recurrence on survival in resected osteosarcoma. Eur J Cancer. 2001 Jan;37(1):39-46. doi: 10.1016/s0959-8049(00)00362-2. PMID 11165128
- [Background] Lucidarme N, Valteau-Couanet D, Oberlin O, Couanet D, Kalifa C, Beaujean F, Lapierre V, Hartmann O. Phase II study of high-dose thiotepa and hematopoietic stem cell transplantation in children with solid tumors. Bone Marrow Transplant. 1998 Sep;22(6):535-40. doi: 10.1038/sj.bmt.1701395. PMID 9758339
- [Background] Hagen B, Walseth F, Walstad RA, Iversen T, Nilsen OG. Single and repeated dose pharmacokinetics of thio-TEPA in patients treated for ovarian carcinoma. Cancer Chemother Pharmacol. 1987;19(2):143-8. doi: 10.1007/BF00254567. PMID 3105905
- [Background] Hart RD, Perloff M, Holland JF. One-day VATH (vinblastine, Adriamycin, thiotepa, and Halotestin) therapy for advanced breast cancer refractory to chemotherapy. Cancer. 1981 Oct 1;48(7):1522-7. doi: 10.1002/1097-0142(19811001)48:73.0.co;2-g. PMID 6793224
- [Background] Heideman RL, Cole DE, Balis F, Sato J, Reaman GH, Packer RJ, Singher LJ, Ettinger LJ, Gillespie A, Sam J, et al. Phase I and pharmacokinetic evaluation of thiotepa in the cerebrospinal fluid and plasma of pediatric patients: evidence for dose-dependent plasma clearance of thiotepa. Cancer Res. 1989 Feb 1;49(3):736-41. PMID 2491958
- [Background] Lazarus HM, Reed MD, Spitzer TR, Rabaa MS, Blumer JL. High-dose i.v. thiotepa and cryopreserved autologous bone marrow transplantation for therapy of refractory cancer. Cancer Treat Rep. 1987 Jul-Aug;71(7-8):689-95. PMID 3111687
- [Background] Kletzel M, Kearns GL, Wells TG, Thompson HC Jr. Pharmacokinetics of high dose thiotepa in children undergoing autologous bone marrow transplantation. Bone Marrow Transplant. 1992 Aug;10(2):171-5. PMID 1525606
- [Background] Kalifa C, Hartmann O, Demeocq F, Vassal G, Couanet D, Terrier-Lacombe MJ, Valteau D, Brugieres L, Lemerle J. High-dose busulfan and thiotepa with autologous bone marrow transplantation in childhood malignant brain tumors: a phase II study. Bone Marrow Transplant. 1992 Apr;9(4):227-33. PMID 1534708
- [Background] Finlay JL, Goldman S, Wong MC, Cairo M, Garvin J, August C, Cohen BH, Stanley P, Zimmerman RA, Bostrom B, Geyer JR, Harris RE, Sanders J, Yates AJ, Boyett JM, Packer RJ. Pilot study of high-dose thiotepa and etoposide with autologous bone marrow rescue in children and young adults with recurrent CNS tumors. The Children's Cancer Group. J Clin Oncol. 1996 Sep;14(9):2495-503. doi: 10.1200/JCO.1996.14.9.2495. PMID 8823328
- [Background] Entz-Werle N, Stoetzel C, Berard-Marec P, Kalifa C, Brugiere L, Pacquement H, Schmitt C, Tabone MD, Gentet JC, Quillet R, Oudet P, Lutz P, Babin-Boilletot A, Gaub MP, Perrin-Schmitt F. Frequent genomic abnormalities at TWIST in human pediatric osteosarcomas. Int J Cancer. 2005 Nov 10;117(3):349-55. doi: 10.1002/ijc.21068. PMID 15900593
- [Background] Bertolini F, Mancuso P, Shaked Y, Kerbel RS. Molecular and cellular biomarkers for angiogenesis in clinical oncology. Drug Discov Today. 2007 Oct;12(19-20):806-12. doi: 10.1016/j.drudis.2007.08.011. Epub 2007 Sep 27. PMID 17933680
- [Background] Oliveira ID, Petrilli AS, Tavela MH, Zago MA, de Toledo SR. TNF-alpha, TNF-beta, IL-6, IL-10, PECAM-1 and the MPO inflammatory gene polymorphisms in osteosarcoma. J Pediatr Hematol Oncol. 2007 May;29(5):293-7. doi: 10.1097/MPH.0b013e3180587e69. PMID 17483704
- [Background] Nardin A, Lefebvre ML, Labroquere K, Faure O, Abastado JP. Liposomal muramyl tripeptide phosphatidylethanolamine: Targeting and activating macrophages for adjuvant treatment of osteosarcoma. Curr Cancer Drug Targets. 2006 Mar;6(2):123-33. doi: 10.2174/156800906776056473. PMID 16529542
- [Background] Entz-Werle N, Schneider A, Kalifa C, Voegeli AC, Tabone MD, Marec-Berard P, Marcellin L, Pacquement H, Terrier P, Boutard P, Meyer N, Gaub MP, Lutz P, Babin A, Oudet P. Genetic alterations in primary osteosarcoma from 54 children and adolescents by targeted allelotyping. Br J Cancer. 2003 Jun 16;88(12):1925-31. doi: 10.1038/sj.bjc.6600968. PMID 12799638
- [Background] Entz-Werle N, Marcellin L, Gaub MP, Guerin E, Schneider A, Berard-Marec P, Kalifa C, Brugiere L, Pacquement H, Schmitt C, Tabone MD, Jeanne-Pasquier C, Terrier P, Dijoud F, Oudet P, Lutz P, Babin-Boilletot A. Prognostic significance of allelic imbalance at the c-kit gene locus and c-kit overexpression by immunohistochemistry in pediatric osteosarcomas. J Clin Oncol. 2005 Apr 1;23(10):2248-55. doi: 10.1200/JCO.2005.03.119. PMID 15800315
- [Background] Freedman LS. Tables of the number of patients required in clinical trials using the logrank test. Stat Med. 1982 Apr-Jun;1(2):121-9. doi: 10.1002/sim.4780010204. PMID 7187087
- [Background] Schemper M, Smith TL. A note on quantifying follow-up in studies of failure time. Control Clin Trials. 1996 Aug;17(4):343-6. doi: 10.1016/0197-2456(96)00075-x. No abstract available. PMID 8889347
- [Background] Rialland F.Treatment and outcome of relapsed osteosarcoma:experience of the societe française des cancers de l'enfant.(in press). 2008. Ref type:in press
- [Background] Sutow WW, Herson J, Perez C. Survival after metastasis in osteosarcoma. Natl Cancer Inst Monogr. 1981 Apr;(56):227-31. PMID 6946292
- [Background] Gelderblom H, Jinks RC, Sydes M, Bramwell VH, van Glabbeke M, Grimer RJ, Hogendoorn PC, McTiernan A, Lewis IJ, Nooij MA, Taminiau AH, Whelan J; European Osteosarcoma Intergroup. Survival after recurrent osteosarcoma: data from 3 European Osteosarcoma Intergroup (EOI) randomized controlled trials. Eur J Cancer. 2011 Apr;47(6):895-902. doi: 10.1016/j.ejca.2010.11.036. Epub 2011 Jan 6. PMID 21216138
- [Background] Leary SE, Wozniak AW, Billups CA, Wu J, McPherson V, Neel MD, Rao BN, Daw NC. Survival of pediatric patients after relapsed osteosarcoma: the St. Jude Children's Research Hospital experience. Cancer. 2013 Jul 15;119(14):2645-53. doi: 10.1002/cncr.28111. Epub 2013 Apr 26. PMID 23625626
- [Background] Beron G, Euler A, winkley K.pulmonary metastase from osteogenic sarcoma: Complete resection and effective chemotherapy contributing to improved prognosis.Eur Paediatr Haematol Oncol 1985; 2:77-85
- [Background] Kaplan EL MP.Nonparametric estimation from incomplete observations.J Am Stat Assoc 1958